CLINICAL TRIAL: NCT01858857
Title: Pharmacovigilance in Gerontopsychiatric Patients
Brief Title: Geriatric Psychiatry and Pharmacovigilance
Acronym: GAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Institut für Arzneimittelsicherheit in der Psychiatrie AMSP e.V. (Unknown); Asklepios Fachklinikum Brandenburg (Unknown); Asklepios Fachklinikum Lübben für Psychiatrie, Psychotherapie und Psychosomatik (Unknown); Asklepios Fachklinikum Teupitz für Psychiatrie (Unknown); Krankenhaus Hedwigshöhe (Unknown); Kompetenznetz TDM KJP e.V. (Unknown)
Responsible Party: Principal Investigator, Helge Frieling,MD, Professor Dr. Helge Frieling, Deputy Director of the Department of psychiatry, social psychiatry and psychotherapy, Hannover Medical School
Other Study IDs: GAP2013; V-15222/68605/2012-2015 (Other Grant/Funding Number: Federal Institute for Drugs and Medical Devices (BfArM))
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Dementia; Depression; Schizophrenia; Psychosomatic Disorders; Anxiety Disorders
Keywords: geriatric psychiatry; pharmacovigilance
MeSH Terms: conditions — Dementia; Depression; Schizophrenia; Psychophysiologic Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Geriatric psychiatric in patients

SUMMARY:
The purpose of this observational multicenter-study is to investigate safety of psychopharmacological treatment and rates of adverse drug reactions in gerontopsychiatric inpatients. Elderly people are at higher risk for developing side effects under pharmacological treatment due to an altered metabolic situation, higher comorbidity rates and often polypharmacy. Furthermore gerontopsychiatric patients can often not articulate their symptoms clearly, for example due to pronounced cognitive impairment.

The aim of the study is to gain valid data of possible adverse drug reaction rates, their potential risk factors and outcome, as well as medical prescription practises.

To assess these outcomes an intensive pharmacovigilance-monitoring will be conducted at the five participating study sites.

At Baseline demographic data, previous and present disorders, use of drugs, previous and present medication, quality of life, cognitive function, physical examination results, laboratory results and ECG will be assessed.

Afterwards patients are visited weekly and screened for possible adverse drug reactions. All adverse drug reactions will be coded in the MedDRA-system.

In case of a possible serious adverse drug reaction serum levels of all psychotropic substances applicated will be assessed. Drug combinations will be analysed using an established advanced bioinformatic tool (mediQ). Diagnosis, medication intake and possible adverse drug reactions are documented continually.

2 weeks after discharge from the ward, patients will be contacted by phone to assess catamnestic data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65+ years old
2. Inpatients treated at one of the geriatric psychiatry study sites.
3. Signed consent form ( Patient and/or legally authorized custodian)

Exclusion Criteria:

1. Patients that are incapable to give their informed consent and are not under legally authorized custodianship.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All inpatients meeting the Inclusion/Exclusion criteria, treated at one of the geriatric psychiatry study sites (one university hospital and four primary care clinics), should be screened.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of frequency and severity of adverse events in geriatric psychiatry inpatients under psychopharmacological treatment | Patients will be monitored continuosly during the hospital stay (expected average of 4 weeks) and at follow-up, which is 2 weeks after discharge.

SECONDARY OUTCOMES:
Assessment of cognitive functioning | At baseline visit and last visit, max. 3 days before discharge from the ward (expected average of hospital stay: 4 weeks).
  Mini Mental State Exam
Quality of life | At baseline visit and last visit, max. 3 days before discharge from the ward (expected average of hospital stay: 4 weeks).
Adverse drug reactions | Patients will be monitored continuosly during the hospital stay (expected average of 4 weeks) and at follow-up, which is 2 weeks after discharge.
Serum levels of substances | 1 day at occurence of SAE
Electrocardiogram | At baseline visit and last visit, max. 3 days before discharge from the ward (expected average of hospital stay: 4 weeks).
Medication intake | Patients medication intake 2 weeks before hospitalisation, continuosly during the hospital stay and at follow-up 2 weeks after discharge will be assessed (expected average of 8 weeks).
  Before hospitalisation and after discharge by interview, during the hospital stay by patients chart.

CONTACTS AND LOCATIONS:
Overall Officials: Helge Frieling, MD, Principal Investigator — MHH; Sermin Toto, MD, Study Director — MHH; Stefan Bleich, MD, Study Chair — MHH
Locations (5):
- Germany (5):
  - Krankenhaus Hedwigshöhe, Berlin
  - Asklepios Fachklinikum Brandenburg, Brandenburg
  - Hannover Medical School, Hanover
  - Asklepios Fachklinikum Lübben, Lubin
  - Asklepios Fachklinikum Teupitz, Teupitz